CLINICAL TRIAL: NCT00998179
Title: Effect of Acu-Transcutaneous Electrical Nerve Stimulation (Acu-TENS) on Post-exercise Expiratory Flow Volume in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Prof. Alice Jones, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: RS9/10
Record Dates: First submitted 2009-10-18; First posted 2009-10-20 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: TENS; acupuncture; FEV1; Normal Healthy subjects

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Acu-TENS (Active Comparator): Application of Acu-TENS prior to exercise
  Interventions: Device: Acu-TENS
- Placebo-TENS (Placebo Comparator): Application of Acu-TENS (without electrical output from the machine) prior to exercise
  Interventions: Device: Placebo-TENS

INTERVENTIONS:
Device: Acu-TENS — Application of Acu-TENS (with electrical output from the machine)
  Arms: Acu-TENS
Device: Placebo-TENS — Application of Acu-TENS (without electrical output from the machine)
  Arms: Placebo-TENS

SUMMARY:
This study aims to investigate the effect of Acu-TENS on forced expiratory volume in one second (FEV1), a test of pulmonary function used to assess airway resistance, during sub-maximal treadmill exercise in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* With normal health

Exclusion Criteria:

* Suffered from respiratory, cardiovascular, musculoskeletal, neurological or endocrine disorders
* No allergic to gel

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)

PRIMARY OUTCOMES:
Forced expiratory flow volume in one second (FEV1)and forced vital capacity (FVC) | before and immediate after the exercise test
Forced expiratory flow volume in one second (FEV1) and forced vital capacity (FVC) | at 15min, 30 min and 45min after the exercise test

SECONDARY OUTCOMES:
Exercise duration | Immediately after the exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Alice Jones, PhD, FACP, Principal Investigator — Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Locations (1):
- Cardiopulmonary and exercise physiology laboratory, The Hong Kong Polytechnic University, Hong Kong, China